CLINICAL TRIAL: NCT02561169
Title: A Randomized Controlled Trial of Oseltamivir in High-Risk Patients Presenting to the Emergency Department With Influenza
Brief Title: A Trial of Oseltamivir in High-Risk Patients Presenting to the Emergency Department With Influenza
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: University of Calgary (Other); University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: Oseltamivir - 2015
Record Dates: First submitted 2015-09-22; First posted 2015-09-25 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Influenza
Keywords: antiviral; oseltamivir
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Oseltamivir (Experimental): 75 mg oseltamivir orally twice daily for 5 days within 72 hours of symptom onset
  Interventions: Drug: Oseltamivir
- Placebo (Placebo Comparator): 75mg placebo calcium carbonate pills taken twice daily for five days within 72 hours of symptom onset and will be identical in appearance to oseltamivir
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Oseltamivir — Those randomized to the intervention will receive oseltamivir 75 mg orally twice daily for 5 days within 72 hours of symptom onset. For patients with a known creatinine clearance < 10 ml/min, the recommended dose of 75mg orally daily for 5 days of either intervention or placebo will be administered.
  Other Names: Tamiflu
  Arms: Oseltamivir
Other: Placebo — Those randomized to the control arm will receive 75mg placebo calcium carbonate pills taken twice daily for five days within 72 hours of symptom onset and will be identical in appearance to oseltamivir. For patients with a known creatinine clearance < 10 ml/min, the recommended dose of 75mg orally daily for 5 days of either intervention or placebo will be administered.
  Other Names: Calcium Carbonate
  Arms: Placebo

SUMMARY:
A multi-centre, randomized, placebo controlled, trial. Participants will be patients either ≥65 years or with one or more high risk conditions presenting to one of four academic emergency departments in Edmonton or Calgary with influenza-like illness. The investigators will test for influenza using a point-of-care rapid test and if positive for influenza participants will be randomized to oseltamivir or placebo and followed prospectively. The primary outcome will be hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient at the University of Alberta Hospital, the Northeast Community Centre, Foothills Medical Centre, Rockyview General Hospital emergency departments
* ≥ 18 years of age
* ≥ 65 years of age OR chronic cardiac or pulmonary disorders (including bronchopulmonary dysplasia, cystic fibrosis, and asthma) , diabetes mellitus and other metabolic diseases, cancer, immunodeficiency, immunosuppression (due to underlying disease and/or therapy), renal disease, anemia, and hemoglobinopathy, any condition that can compromise respiratory function or the handling of respiratory secretions or that can increase the risk of aspiration
* Acute respiratory infection (ARI) exhibiting 2 or more symptoms, onset within last 72 hours
* Laboratory confirmation of influenza infection, onset within last 72 hours

Exclusion Criteria:

* Contraindication to oseltamivir (i.e., previous anaphylaxis)
* Resident of a nursing home
* Canadian Triage and Acuity Scale (CTAS) 1
* Blood pressure < 90 mmHg
* Respiratory rate >30 breaths per minute
* PaO2 less <88%
* Confusion
* Inability to eat or drink
* Radiographic evidence of pneumonia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Non-elective Hospitalizations (number of hospitalizations) | 28 days
Length of non-elective hospitalization (days) | 28 days

SECONDARY OUTCOMES:
Lower respiratory tract infection (LRTI), (number of LRTIs) | 28 days
Pneumonia (number of episodes of pneumonia) | 28 days
Acute Sinusitis (number of episodes of acute sinusitis) | 28 Days
New antimicrobial prescription (number of antimicrobial prescriptions) | 28 Days
Medical visits for acute respiratory illness (number of medical visits) | 28 Days
Death | 3 months
Adverse Events (number of adverse events) | 5 days
Admission to intensive or critical care unit (number of admissions) | 28 days
Duration of stay in intensive or critical care unit (days) | 28 days
Need for mechanical ventilation (number of mechanical ventilation) | 28 days
Duration of mechanical ventilation (days) | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Mark Loeb, MD, Principal Investigator — McMaster University
Locations (1):
- Foothills Medical Centre Emergency Department, Calgary, Alberta, Canada